CLINICAL TRIAL: NCT03639415
Title: Phase II Study of Change the Dose Frequency of Controlled-Release Oxycodone to Refractory Pain
Brief Title: Change the Dose Frequency of Controlled-Release Oxycodone to Refractory Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: There is no fund to support
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF010
Record Dates: First submitted 2018-06-28; First posted 2018-08-21 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2018-06

CONDITIONS: Cancer Pains
Keywords: Opioid; Refractory Pain; dose frequency; nausea; vomit; dizziness
MeSH Terms: conditions — Cancer Pain; Pain, Intractable; Nausea; Vomiting; Dizziness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- controlled-release oxycodone group (Experimental): Patients with moderate to severe pain accept CR oxycodone treatment and if any follow situations appears, then change the dose frequency from every 12 hours to every 8 hours or 6 hours.
  1. Patients are satisfied with the pain control, but unable to tolerate nausea、vomit or dizziness, and can't get satisfactory pain control if reducing the CR oxycodone dose.
  2. Patients are unsatisfied with the pain control, but can't increase the CR oxycodone dose because of intolerable nausea、vomit or dizziness.
  Interventions: Drug: Increasing the Controlled-Release Oxycodone dose frequency

INTERVENTIONS:
Drug: Increasing the Controlled-Release Oxycodone dose frequency — Keep the daily dose while increase the dose frequency of Controlled-Release Oxycodone so that reduce the single dose

SUMMARY:
Many patients with cancer experience moderate to severe pain that requires treatment with strong opioids, of which oxycodone and morphine are examples, they are widely applied in clinical treatment because of sustained-released formulation can reduce dosing frequency. Goal of pain management is get adequate analgesia and minimize the adverse event at the same time, but in fact there are about 10%-30% patients can't get adequate analgesia because of intolerable adverse event. The common adverse event of Controlled-Release Oxycodone(CR Oxycodone ) are nausea (29.9%)、constipation （25.4%）、dizziness（22.4%） and vomit（11.9%），about 32.8% patients treatment was discontinued because of these adverse event. The peak concentration of opioid is related to adverse event, while the valley concentration is correlated to the analgesic effect. Therefore, if we keep the daily dose while increase the dose frequency so that reduce the single dose, it's will help to avoid intolerable adverse event caused by excessive opioid peak concentration and keep the opioid analgesia at the same time. It's a reasonable way to solve the side effects of opioid.

In order to explore the effect of change the dosing frequency of CR Oxycodone to treat refractory pain, pre-experiment have done by several clinical centrals in Fujian province. Preliminary results show that for the patients who can't accept the current opioid dose because of intolerable side effect, changing the dosing frequency is a safe and effect way.

DETAILED DESCRIPTION:
This is a multicenter、singe arm、prospective study.

Study population:

Moderate to severe cancer pain (4-6 on the standard Numerical Rating Scale [NRS], range 0-10) patients with unsatisfactory pain control because of intolerable nausea、vomit or dizziness during accept CR Oxycodone treatment.

Therapeutic schemes:

1. CR oxycodone dose titration scheme: adjusting the dose of CR oxycodone every 24 hours according to the NRS and adverse event;
2. Increasing the dose frequency scheme; Patients with moderate to severe pain accept CR oxycodone treatment and if any follow situations appears, then change the dose frequency from every 12 hours to every 8 hours or 6 hours.

Patients are satisfied with the pain control, but unable to tolerate nausea、vomit or dizziness, and can't get satisfactory pain control if reducing the CR oxycodone dose.

Patients are unsatisfied with the pain control, but can't increase the CR oxycodone dose because of intolerable nausea、vomit or dizziness.

Primary end point:

The effective rate of treatment: the rate of patients who get satisfactory pain control without intolerable adverse event in two consecutive day .

Secondary end point:

The time of reach effective treatment； The degree of pain reduction; The incident rate of adverse drug reaction The reduction rate of adverse drug reaction The change of plasm concentration after change the dose frequency; The relationship between peripheral blood gene and analgesia effect; The relationship between peripheral blood gene and adverse event;

ELIGIBILITY:
Inclusion Criteria:

* Opioid naïve or tolerate patients with moderate to severe cancer pain (NRS≥4). Opioid naïve includes patients who are not chronically receiving opioid analgesic on a daily basis and therefore have not developed significant tolerance. The FDA identifies tolerance as receiving at least 60 mg of morphine daily, at least 30 mg of oral oxycodone daily, or at least 8 mg of oral hydromorphone daily or an equianalgesic dose of another opioid for a week or longer.
* Age≥18 years old
* The effect of antitumor therapy (radiotherapy, chemotherapy, targeted therapy, etc.) on analgesia can be excluded during the period of analgesic drug dose adjustments
* Patients can well communicate and cooperate with doctors, understand the therapeutic schemes, agree to attend the study and signed the informed consent form.

Exclusion Criteria:

* Allergic to research drugs
* Pain of noncancerous or unknown cause, such as osteoarthritis pain, low back pain, etc.
* Acute pain
* Patients receiving radiotherapy or chemotherapy during the period of the treatment
* No defecation in the first 3 days before enrollment
* Patients with opioid contraindication: Respiratory inhibition; head damage; paralytic bowel obstruction; acute abdomen; chronic obstructive airway disease; pulmonary heart disease; chronic bronchial asthma; hypercapnia.
* Use of monoamine oxidase inhibitors within 1 week before enrollment
* Abnormal laboratory indexes with obvious clinical significance： creatinine beyond two times of the upper limit of normal value;ALT or AST beyond 2.5 times of the upper limit of normal value (For patients with liver metastasis, ALT or AST beyond 5 times of the upper limit of normal value); Liver function Child grade C
* Acute abdominal disease or accept surgical procedures which may cause gastrointestinal stricture, blind loop or gastrointestinal obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
The effective rate of treatment | 2 years
  At study entry, assess the adverse drug reaction (ADR) and the pain degree by Likert scale everyday. The Likert scale of pain includes the absence of pain (a score of 0), mild pain (a score of 1), moderate pain (a score of 2), severe pain (a score of 3). The Likert scale of ADR includes the absence of ADR (a score of 0), mild ADR (a score of 1), moderate ADR (a score of 2), severe ADR (a score of 3).
  The effective rate of treatment: the rate of patients who get satisfactory pain control (0 or 1 point on the 3-point Likert scale ) without intolerable adverse event (0 or 1 point on the 3-point Likert scale ) in two consecutive day .

SECONDARY OUTCOMES:
The time of reach effective treatment | 2 years
  Effective treatment means patients who get satisfactory pain control (0 or 1 point on the 3-point Likert scale ) without intolerable adverse event (0 or 1 point on the 3-point Likert scale ) in two consecutive day .
The degree of pain reduction | 2 years
  Apply the Likert scale to evaluate pain degree. The Likert scale of pain includes the absence of pain (a score of 0), mild pain (a score of 1), moderate pain (a score of 2), severe pain (a score of 3).
The incident rate of adverse drug reaction | 2 years
The reduction rate of adverse drug reaction | 2 years
Oxycodone blood concentration monitoring | 2 years
  The blood samples are collected before and after changing the oxycodone dose frequency，For the patients whose frequency change from every 12 hours to every 8 hours ,the blood sampling time points are one hour before changing dose and one hour ,four hour after changing dose, For the patients whose frequency change from every 12 hours to every 6 hours ,the blood sampling time points are one hour before changing dose and one hour ,three hour after changing dose
Detection of patient's peripheral blood gene | 2 years
  The blood samples are collected before change the oxycodone dose frequency, and apply the Next-generation sequencing technology to check patient's peripheral blood geneblood gene

IPD SHARING:
Plan to Share IPD: No